CLINICAL TRIAL: NCT00654810
Title: Exercise Rehabilitation of Younger and Older People With Claudication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Andrew W. Gardner, PhD, University of Oklahoma Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0097; K01AG000657 (NIH)
Record Dates: First submitted 2008-04-07; First posted 2008-04-09 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2008-04

CONDITIONS: Intermittent Claudication
Keywords: functional ability; gait; musculoskeletal disorder therapy; peripheral blood vessel disorder
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Low intensity group (40% of maximal exercise capacity)
  Interventions: Behavioral: Walking Exercise
- 2 (Experimental): High intensity group (80% of maximal exercise capacity)
  Interventions: Behavioral: Walking Exercise

INTERVENTIONS:
Behavioral: Walking Exercise — Intermittent treadmill walking to near maximal claudication pain three days per week

SUMMARY:
The purpose of this study is to examine the effect of age and the effect of exercise intensity of rehabilitation programs on claudication pain symptoms and leg circulation of younger and older patients with intermittent claudication.

DETAILED DESCRIPTION:
Thirty-one patients randomized to low-intensity exercise rehabilitation and 33 patients randomized to high-intensity exercise rehabilitation completed the study. The 6-month exercise rehabilitation programs consisted of intermittent treadmill walking to near maximal claudication pain three days per week at either 40% (low-intensity group) or 80% (high-intensity group) of maximal exercise capacity. Total work performed in the two training regimens was similar by having the patients in the low-intensity group exercise for a longer duration than patients in the high-intensity group. Measurements of physical function, peripheral circulation, and health-related quality of life were obtained on each patient before and after the rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* History of intermittent claudication
* Exercise tolerance limited by intermittent claudication during a screening treadmill test
* Ankle/brachial index (ABI) at rest less than 0.90
* Live independently at home

Exclusion Criteria:

* Absence of PAD (peripheral artery disease)
* Asymptomatic PAD (Fontaine stage I)
* Rest pain PAD (Fontaine stage III)
* Exercise tolerance limited by factors other than claudication (e.g., coronary artery disease, dyspnea, poorly controlled blood pressure)
* Active cancer, renal disease, or liver disease
* Current use of pentoxifylline or cilostazol medications for the treatment of intermittent claudication

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 1994-02; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
Change in the walking distance to onset of leg pain, and the change in walking distance to maximal leg pain. | 6 months

SECONDARY OUTCOMES:
Changes in cardiopulmonary function, calf muscle circulation, and health-related quality of life. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W. Gardner, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Gardner AW, Poehlman ET. Exercise rehabilitation programs for the treatment of claudication pain. A meta-analysis. JAMA. 1995 Sep 27;274(12):975-80. PMID 7674529
- [Background] Gardner AW, Katzel LI, Sorkin JD, Bradham DD, Hochberg MC, Flinn WR, Goldberg AP. Exercise rehabilitation improves functional outcomes and peripheral circulation in patients with intermittent claudication: a randomized controlled trial. J Am Geriatr Soc. 2001 Jun;49(6):755-62. doi: 10.1046/j.1532-5415.2001.49152.x. PMID 11454114
- [Background] Gardner AW, Katzel LI, Sorkin JD, Goldberg AP. Effects of long-term exercise rehabilitation on claudication distances in patients with peripheral arterial disease: a randomized controlled trial. J Cardiopulm Rehabil. 2002 May-Jun;22(3):192-8. doi: 10.1097/00008483-200205000-00011. PMID 12042688
- [Background] Gardner AW, Killewich LA, Montgomery PS, Katzel LI. Response to exercise rehabilitation in smoking and nonsmoking patients with intermittent claudication. J Vasc Surg. 2004 Mar;39(3):531-8. doi: 10.1016/j.jvs.2003.08.037. PMID 14981444
- [Result] Gardner AW, Montgomery PS, Flinn WR, Katzel LI. The effect of exercise intensity on the response to exercise rehabilitation in patients with intermittent claudication. J Vasc Surg. 2005 Oct;42(4):702-9. doi: 10.1016/j.jvs.2005.05.049. PMID 16242558
- [Result] Gardner AW, Katzel LI, Sorkin JD, Killewich LA, Ryan A, Flinn WR, Goldberg AP. Improved functional outcomes following exercise rehabilitation in patients with intermittent claudication. J Gerontol A Biol Sci Med Sci. 2000 Oct;55(10):M570-7. doi: 10.1093/gerona/55.10.m570. PMID 11034229
- [Derived] Gardner AW, Montgomery PS, Parker DE. Optimal exercise program length for patients with claudication. J Vasc Surg. 2012 May;55(5):1346-54. doi: 10.1016/j.jvs.2011.11.123. Epub 2012 Mar 28. PMID 22459748